CLINICAL TRIAL: NCT03370289
Title: An Open-label Phase 4 Study to Evaluate the Immunogenicity and Safety of Intramuscular Injections of BLB-750 in Healthy Adult Subjects
Brief Title: A Phase 4 Post-marketing Study of Intramuscular Injections of BLB-750 in Healthy Adult Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BLB-750/CCT-901; U1111-1198-2695 (Other: WHO); JapicCTI-173797 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2017-12-07; First posted 2017-12-12 (Actual); Results first posted 2019-07-29 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-06

CONDITIONS: Pandemic Influenza Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BLB-750 Qinghai RG strain (Experimental): Two doses of BLB-750 Qinghai reverse genetics (RG) strain at a vaccination dose of 0.5 mL (HA antigen level of 7.5 µg per strain) will be injected into the upper arm muscle (the deltoid muscle) at 3-week intervals (Day 1 and Day 22) in a treatment period of 43 days.
  Interventions: Biological: BLB-750 Vaccine (Qinghai RG strain)

INTERVENTIONS:
Biological: BLB-750 Vaccine (Qinghai RG strain) — BLB-750 Injection
  Other Names: Cell-Culture Influenza Vaccine H5N1 "Takeda"

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of two intramuscular vaccinations with BLB-750 in healthy Japanese adults.

DETAILED DESCRIPTION:
The drug being tested in this study is called BLB-750 that is a vaccine for pandemic influenza infection. This study will evaluate immunogenicity and safety of two intramuscular vaccinations with BLB-750 at 3-week intervals in healthy Japanese adults. The study will enroll 55 participants. BLB-750 will be administered in opened manner:

- Two intramuscular vaccinations of BLB-750 at 3-week intervals, 0.5 mL

This trial will be conducted in Japan. The overall time to participate in this study will be 43 days, starting on the day of first vaccination. Participants will make multiple visits to the clinic, including 21 days after the first vaccination and 21 days after the second vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant signs and dates a written, informed consent form prior to the initiation of any study procedures.
3. The participant is a healthy Japanese adult man or woman.
4. The participant is aged 20 to 49 years, inclusive, at the time of informed consent.
5. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study.

Exclusion Criteria:

1. The participant has received vaccination with any other investigational products within 4 months prior to vaccination with the study drug.
2. The participant has a history of vaccination with an H5N1 influenza vaccine.
3. The participant has a history of infection with H5N1 virus.
4. The participant is at high risk of contracting H5N1 influenza infection (e.g., poultry workers).
5. The participant is an immediate family member, study site employee, or is in a dependant relationship with a study site employee who is involved in conduct of this study (e.g., spouse, parent, child, sibling) or may consent under duress.
6. The participant has poorly controlled, clinically significant manifestations of neurological, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, endocrine, or other disorders, which may impact their ability to participate as participants or may potentially confound the study results.
7. The participant has a body temperature (oral) ≥37.5°C prior to vaccination with the study drug on Day 1.
8. The participant has any medically diagnosed or suspected immune-deficiency condition.
9. The participant has an immunocompromising condition or disease, or is currently undergoing a form of treatment or was undergoing a form of treatment that can be expected to influence immune response within 30 days prior to vaccination with the study drug.

   Such treatments include, but are not limited to, systemic or high dose inhaled corticosteroids (>800 μg/day of beclomethasone dipropionate or equivalent; the use of inhaled and nasal steroids that do not exceed this level will be permitted), radiation treatment or other immunosuppressive or cytotoxic drugs.
10. The participant has received antipyretics within 4 hours prior to vaccination with the study drug.
11. The participant has a history of Guillain-Barré Syndrome, demyelinating disorders (including acute disseminated encephalomyelitis [ADEM] and multiple sclerosis), or convulsions.
12. The participant has a functional or anatomic asplenia.
13. The participant has a rash, other dermatologic conditions or tattoos that may interfere with the evaluation of local reaction.
14. The participant has a past or present history of infection with the Hepatitis B Virus (HBV), Hepatitis C Virus (HCV) or Human Immunodeficiency Virus (HIV).
15. The participant has a known hypersensitivity to any component of BLB-750.
16. The participant has a history of severe allergic reactions or anaphylaxis.
17. The participant has a history of drug abuse (defined as any illicit drug use) or a history of alcohol dependence within 1 year prior to vaccination with the study drug or is unwilling to agree to abstain from excessive alcohol and drugs throughout the study.
18. The participant has received any blood product (e.g., blood transfusion or immunoglobulin) within 90 days prior to vaccination with the study drug.
19. The participant has received any live vaccine within 4 weeks (28 days) prior to vaccination with the study drug or any inactivated vaccine within 2 weeks (14 days) prior to vaccination with the study drug.
20. The participant is a pregnant or lactating woman or wishes to become pregnant before signing informed consent, during, or within 12 weeks after the last vaccination with the study drug or intends to donate ova during such time period.
21. For males: The participant has donated whole blood ≥200 mL within 4 weeks (28 days) or ≥400 mL within 12 weeks (84 days) prior to the first vaccination with the study drug.

    For females: The participant has donated whole blood ≥200 mL within 4 weeks (28 days) or ≥400 mL within 16 weeks (112 days) prior to the first vaccination with the study drug.
22. For males: The participant has donated whole blood ≥800 mL in total within 52 weeks (364 days) prior to the first vaccination with the study drug.

    For females: The participant has donated whole blood ≥400 mL in total within 52 weeks (364 days) prior to the first vaccination with the study drug.
23. The participant has donated blood components within 2 weeks (14 days) prior to the first vaccination with the study drug.
24. In the opinion of the investigator, the participant is unlikely to comply with protocol requirements or is considered ineligible for any other reason.
25. The participant has presence of thrombocytopenia or coagulopathy, or has received anticoagulant therapy within 30 days prior to the first vaccination with the study drug.

Ages: 20 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Sekino Rinsho Yakuri Clinic, Toshima-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at one investigative site in Japan, from 12 January 2018 to 28 February 2018.
Pre-assignment Details: Healthy volunteer were enrolled and vaccinated the study drug, BLB-750 at a 3-week interval (Day 1 and Day 22) in a treatment period of 43 days through intramuscular route.
Groups:
- Overall (BLB-750 Vaccine): Two doses of BLB-750 Qinghai reverse genetics (RG) strain at a vaccination dose of 0.5 mL (HA antigen level of 7.5 μg per strain) were injected into the upper arm muscle (the deltoid muscle) at 3-week intervals (Day 1 and Day 22) in a treatment period of 43 days.
Period: Overall Study
Arm/Group | Overall (BLB-750 Vaccine)
Started | 55
Completed | 50
Not Completed | 5
Not completed — Screen Failure | 1
Not completed — Sample Size Sufficient | 4

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All participants who received at least 1 dose of the study drug for the treatment period.
Arm/Group | Overall (BLB-750 Vaccine)
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.3 (4.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  Japan | 55
Height [Mean (Standard Deviation); unit: Centimeter (cm)] | 165.5 (9.06)
Weight [Mean (Standard Deviation); unit: Kilogram (kg)] | 58.43 (7.567)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — Body Mass Index = weight (kg)/[height (m)^2]
  kilogram per square meter (kg/m^2) | 21.29 (1.657)
Single Radial Hemolysis (SRH) Antibody Titer [Mean (Standard Deviation); unit: mm^2] | 4.0 (0.00)
Number of Participants who Had No Infection of Influenza within 1 Year prior to Study Start [Count of Participants; unit: Participants] | 55

OUTCOME MEASURES:

1. Primary Outcome: Seroprotection Rate as Measured by Single Radial Hemolysis (SRH) Antibody Titer for the Vaccine Strain at 21 Days After the Second Vaccination
Description: Seroprotection rate was measured by SRH antibody titer for BLB-750 Qinghai RG strain at 21 days after second vaccination. Seroprotection rate as SRH antibody titer is defined as the percentage of participants with SRH antibody titer ≥25 mm^2.
Time Frame: Day 43 (21 days after the second vaccination)
Population: Full Analysis Set (FAS): All participants who received at least 1 dose of the study drug for the treatment period.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Overall (BLB-750 Vaccine)
Number analyzed (Participants) | 55
Percentage of participants | 32.7 [20.681 to 46.707]

2. Primary Outcome: Seroconversion Rate as Measured by SRH Antibody Titer for the Vaccine Strain at 21 Days After the Second Vaccination
Description: Seroconversion rate was measured by SRH antibody titer for BLB-750 Qinghai RG strain at 21 days after second vaccination. Seroconversion rate as SRH antibody titer is defined as the percentage of participants with a 50% or more increase in SRH antibody titer from baseline for those who have a baseline value >4 mm^2 or SRH antibody titer ≥25 mm^2 for those who have a baseline value ≤4 mm^2.
Time Frame: Day 43 (21 days after the second vaccination)
Population: Full Analysis Set (FAS): All participants who received at least 1 dose of the study drug for the treatment period.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Overall (BLB-750 Vaccine)
Number analyzed (Participants) | 55
Percentage of participants | 32.7 [20.681 to 46.707]

3. Primary Outcome: Geometric Mean Fold Increase (GMFI) in SRH Antibody Titer From Baseline for the Vaccine Strain at 21 Days After the Second Vaccination
Description: GMFI was measured as geometric mean fold change from baseline in SRH antibody titer for BLB-750 Qinghai RG strain at 21 days after second vaccination.
Time Frame: Day 43 (21 days after the second vaccination)
Population: Full Analysis Set (FAS): All participants who received at least 1 dose of the study drug for the treatment period.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | Overall (BLB-750 Vaccine)
Number analyzed (Participants) | 55
Fold change | 3.5636 [2.88968 to 4.39463]

4. Secondary Outcome: Seroprotection Rate as Measured by SRH Antibody Titer for the Vaccine Strain at 21 Days After the First Vaccination
Description: Seroprotection rate was measured by SRH antibody titer for BLB-750 Qinghai RG strain at 21 days after first vaccination. Seroprotection rate as SRH antibody titer is defined as the percentage of participants with SRH antibody titer ≥25 mm^2.
Time Frame: Day 22 (21 days after the first vaccination)
Population: Full Analysis Set (FAS): All participants who received at least 1 dose of the study drug for the treatment period.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Overall (BLB-750 Vaccine)
Number analyzed (Participants) | 55
Percentage of participants | 10.9 [4.110 to 22.247]

5. Secondary Outcome: Seroconversion Rate as Measured by SRH Antibody Titer for the Vaccine Strain at 21 Days After the First Vaccination
Description: Seroconversion rate was measured by SRH antibody titer for BLB-750 Qinghai RG strain at 21 days after first vaccination. Seroconversion rate as SRH antibody titer is defined as the percentage of participants with a 50% or more increase in SRH antibody titer from baseline for those who have a baseline value >4 mm^2 or SRH antibody titer ≥25 mm^2 for those who have a baseline value ≤4 mm^2.
Time Frame: Day 22 (21 days after the first vaccination)
Population: Full Analysis Set (FAS): All participants who received at least 1 dose of the study drug for the treatment period.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Overall (BLB-750 Vaccine)
Number analyzed (Participants) | 55
Percentage of participants | 10.9 [4.110 to 22.247]

6. Secondary Outcome: GMFI in SRH Antibody Titer From Baseline for the Vaccine Strain at 21 Days After the First Vaccination
Description: GMFI was measured as geometric mean fold change from baseline in SRH antibody titer for BLB-750 Qinghai RG strain at 21 days after first vaccination.
Time Frame: Day 22 (21 days after the first vaccination)
Population: Full Analysis Set (FAS): All participants who received at least 1 dose of the study drug for the treatment period.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | Overall (BLB-750 Vaccine)
Number analyzed (Participants) | 55
Fold change | 2.3319 [1.87559 to 2.89931]

7. Secondary Outcome: Geometric Mean Titer (GMT) of SRH Antibody Titer for the Vaccine Strain at 21 Days After Each Vaccination
Description: GMT was measured by SRH antibody titer for BLB-750 Qinghai RG strain at 21 days after first and second vaccination.
Time Frame: Day 22, and Day 43 (21 days after the first and the second vaccination)
Population: Full Analysis Set (FAS): All participants who received at least 1 dose of the study drug for the treatment period.
Measure: Geometric Mean (95% Confidence Interval); unit: mm^2
Arm/Group | Overall (BLB-750 Vaccine)
Number analyzed (Participants) | 55
mm^2
  Day 22 | 9.3277 [7.50234 to 11.59725]
  Day 43 | 14.2543 [11.55870 to 17.57854]

8. Secondary Outcome: Number of Participants Reporting Who Had One or More Treatment-emergent Adverse Event (TEAE)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: Up to Day 43
Population: Safety Analysis Set (SAS): All participants who received at least 1 dose of the study drug for the treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Overall (BLB-750 Vaccine)
Number analyzed (Participants) | 55
Participants | 25

9. Secondary Outcome: Number of Participants With Adverse Events Related to Solicited Local and Systemic Adverse Events to be Recorded in the Participant Diary
Description: Local reactions and systemic events were recorded using a diary.
Time Frame: Up to Day 43
Population: Safety Analysis Set (SAS): All participants who received at least 1 dose of the study drug for the treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Overall (BLB-750 Vaccine)
Number analyzed (Participants) | 55
Participants | 24

10. Secondary Outcome: Change From Baseline in Mean Systolic Blood Pressure at Specific Time Points After Vaccination
Time Frame: Baseline, At 30 minutes after the first vaccination and on Day 22 after the first vaccination, and at 30 minutes after the second vaccination and on Day 22 after the second vaccination
Population: Safety Analysis Set (SAS): All participants who received at least 1 dose of the study drug for the treatment period.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Overall (BLB-750 Vaccine)
Number analyzed (Participants) | 55
mmHg
  At 30 Minutes after the 1st Vaccination | -2.2 (8.57)
  Day 22 after the 1st Vaccination | 3.2 (10.73)
  At 30 Minutes after the 2nd Vaccination | -3.3 (11.19)
  Day 22 after the 2nd vaccination | -4.2 (11.06)

11. Secondary Outcome: Change From Baseline in Mean Diastolic Blood Pressure at Specific Time Points After Vaccination
Time Frame: as for outcome 10
Population: Safety Analysis Set (SAS): All participants who received at least 1 dose of the study drug for the treatment period.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Overall (BLB-750 Vaccine)
Number analyzed (Participants) | 55
mmHg
  At 30 Minutes after the 1st Vaccination | -1.0 (6.59)
  Day 22 after the 1st Vaccination | 0.4 (11.53)
  At 30 Minutes after the 2nd Vaccination | 0.0 (9.81)
  Day 22 after the 2nd vaccination | -0.7 (11.89)

12. Secondary Outcome: Change From Baseline in Mean Pulse Rate at Specific Time Points After Vaccination
Time Frame: At 30 minutes after the first vaccination and on Day 22 after the first vaccination, and at 30 minutes after the second vaccination and on Day 22 after the second vaccination
Population: Safety Analysis Set (SAS): All participants who received at least 1 dose of the study drug for the treatment period.
Measure: Mean (Standard Deviation); unit: Beats per minutes
Arm/Group | Overall (BLB-750 Vaccine)
Number analyzed (Participants) | 55
Beats per minutes
  At 30 Minutes after the 1st Vaccination | -4.7 (6.54)
  Day 22 after the 1st Vaccination | 5.5 (9.96)
  At 30 Minutes after the 2nd Vaccination | -8.6 (7.20)
  Day 22 after the 2nd vaccination | -0.4 (8.49)

13. Secondary Outcome: Change From Baseline in Mean Respiratory Rate at 30 Minutes After Vaccination
Time Frame: Baseline, At 30 minutes after the first vaccination, and at 30 minutes after the second vaccination
Population: Safety Analysis Set (SAS): All participants who received at least 1 dose of the study drug for the treatment period.
Measure: Mean (Standard Deviation); unit: Breaths per minutes
Arm/Group | Overall (BLB-750 Vaccine)
Number analyzed (Participants) | 55
Breaths per minutes
  At 30 Minutes after the 1st Vaccination | -0.6 (1.38)
  At 30 Minutes after the 2nd Vaccination | -0.7 (1.72)

14. Secondary Outcome: Mean Body Temperature at Specific Time Points After Vaccination
Time Frame: Baseline, Days 1, 2, 3, 4, 5, 6, 7, and 22 after the first vaccination, Days 1, 2, 3, 4, 5, 6, 7, and 22 after the second vaccination
Population: Safety Analysis Set (SAS): All participants who received at least 1 dose of the study drug for the treatment period.
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | Overall (BLB-750 Vaccine)
Number analyzed (Participants) | 55
degree Celsius
  Day 1 after the 1st Vaccination | 36.70 (0.356)
  Day 2 after the 1st Vaccination | 36.65 (0.324)
  Day 3 after the 1st Vaccination | 36.73 (0.329)
  Day 4 after the 1st Vaccination | 36.64 (0.397)
  Day 5 after the 1st Vaccination | 36.71 (0.293)
  Day 6 after the 1st Vaccination | 36.65 (0.351)
  Day 7 after the 1st Vaccination | 36.69 (0.288)
  Day 1 after the 2nd Vaccination | 36.70 (0.363)
  Day 2 after the 2nd Vaccination | 36.65 (0.322)
  Day 3 after the 2nd Vaccination | 36.65 (0.377)
  Day 4 after the 2nd Vaccination | 36.64 (0.374)
  Day 5 after the 2nd Vaccination | 36.60 (0.403)
  Day 6 after the 2nd Vaccination | 36.72 (0.361)
  Day 7 after the 2nd Vaccination | 36.67 (0.304)

ADVERSE EVENTS:
Time Frame: Up to Day 43
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Overall (BLB-750 Vaccine)
All-Cause Mortality (participants affected / at risk) | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55
Other Adverse Events (participants affected / at risk) | 25/55
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall (BLB-750 Vaccine) (N=55)
Abdominal pain (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Malaise (General disorders) | 12
Fatigue (General disorders) | 9
Injection site pain (General disorders) | 8
Chills (General disorders) | 3
Injection site pruritus (General disorders) | 2
Pyrexia (General disorders) | 2
Injection site erythema (General disorders) | 1
Injection site warmth (General disorders) | 1
Influenza (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 6
Dizziness (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2017-11-21): https://cdn.clinicaltrials.gov/large-docs/89/NCT03370289/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-03): https://cdn.clinicaltrials.gov/large-docs/89/NCT03370289/SAP_001.pdf